CLINICAL TRIAL: NCT00238199
Title: Phase II Study of Calcitriol-Enhanced Docetaxel in Patients With Previously Untreated Metastatic or Locally Advanced Pancreatic Cancer
Brief Title: Calcitriol and Docetaxel in Treating Patients With Metastatic or Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Charles Blanke, Oregon Health and Science University Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445077; OHSU-GIM-02007-L; OHSU-1104
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Calcitriol; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: docetaxel

SUMMARY:
RATIONALE: Calcitriol may cause pancreatic cancer cells to look more like normal cells, and to grow and spread more slowly. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Calcitriol may also help docetaxel work better by making the tumor cells more sensitive to the drug. Giving calcitriol together with docetaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving calcitriol together with docetaxel works in treating patients with metastatic or locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with metastatic or locally advanced pancreatic cancer treated with calcitriol and docetaxel.

Secondary

* Determine the median and one-year survival of patients treated with this regimen.
* Determine the overall response in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the change in pancreatic cancer-induced pain in patients treated with this regimen.

OUTLINE: Patients receive oral calcitriol on days 1, 8, and 15 and docetaxel IV over 15-30 minutes on days 2, 9, and 16. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of pancreatic cancer

  * Locally advanced or metastatic disease

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* Not specified

Hematopoietic

* White blood cell (WBC) > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase (AP) < 5.0 times ULN
* Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) < 2.5 times ULN (if AP < 2.5 times ULN) OR
* ALT and AST < 1.5 times ULN (if AP > 2.5 times ULN and < 5.0 times ULN)

Renal

* Creatinine < 1.3 mg/dL
* Calcium < 10.5 mg/dL
* Phosphate < 4.7 mg/dL
* No kidney stones within the past 5 years
* No history of hypercalcemia

Cardiovascular

* No myocardial infarction within the past 3 months
* No uncontrolled heart failure with a known ejection fraction < 30%
* No other significant heart disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No hypersensitivity to docetaxel or other drugs formulated with polysorbate 80
* No peripheral neuropathy ≥ grade 2
* No comorbid condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for metastatic disease
* No prior chemoradiotherapy for locally advanced disease
* No prior adjuvant docetaxel

  * Other prior adjuvant chemotherapy allowed

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* More than 2 weeks since prior radiotherapy

Surgery

* More than 30 days since prior investigational surgery

Other

* More than 7 days since prior and no concurrent digoxin or thiazide diuretic therapy
* More than 30 days since prior investigational therapy
* No concurrent magnesium-containing antacids, bile resin-binding drugs, or calcium supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Time to progression

SECONDARY OUTCOMES:
Median and one-year survival
Overall response
Toxicity
Change in pancreatic cancer-induced pain

CONTACTS AND LOCATIONS:
Overall Officials: Charles D. Blanke, MD, FACP, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Oregon Health & Science University Cancer Institute, Portland, Oregon, United States